CLINICAL TRIAL: NCT01168687
Title: Placebo-Controlled Crossover Trial of Levetiracetam on Ethanol Intake
Brief Title: Effects of Levetiracetam (Keppra) on Alcohol Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); University of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: H1815-29512-02; W81XWH-05-1-0215 (Other Grant/Funding Number: US Dept. of the Army)
Record Dates: First submitted 2008-10-06; First posted 2010-07-23 (Estimated); Results first posted 2013-02-25 (Estimated); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Alcohol Abuse; Drug Abuse
Keywords: keppra; levetiracetam; alcoholism; genetics; subjective report
MeSH Terms: conditions — Alcoholism; Substance-Related Disorders | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Twenty moderate to heavy social alcohol users will receive 250 mg of levetiracetam BID (500 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 500 mg of levetiracetam BID (1,000 mg/day) x 7 days.
  Interventions: Drug: Levetiracetam (Keppra); Drug: Placebo
- Group B (Experimental): Twenty moderate to heavy social alcohol users will receive 500 mg levetiracetam BID (1000 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 1000 mg levetiracetam BID (2,000 mg per day) x 7 days.
  Interventions: Drug: Levetiracetam (Keppra); Drug: Placebo

INTERVENTIONS:
Drug: Levetiracetam (Keppra) — Group A: Twenty moderate to heavy social alcohol users will receive 250 mg of levetiracetam BID (500 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 500 mg of levetiracetam BID (1,000 mg/day) x 7 days.
  Group B: Twenty moderate to heavy social alcohol users will receive 500 mg levetiracetam BID (1000 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 1000 mg levetiracetam BID (2,000 mg per day) x 7 days.
  Other Names: Keppra
Drug: Placebo

SUMMARY:
The overall goals of this study are to (1) expand knowledge about interactions of levetiracetam with alcohol by assessing the effects of levetiracetam compared to placebo in moderate and heavy social alcohol users and (2) to test the AccuswayTM platform as a tool to measure postural control (which has been used as a marker of intoxication) and the effects of levetiracetam on postural control.

DETAILED DESCRIPTION:
The investigators propose a 42-day, double-blind, placebo-controlled crossover study in light to moderate and heavy alcohol users who are social drinkers.

The specific aims are to:

1. Determine if levetiracetam alters daily alcohol consumption by comparing the mean drinks consumed per day during levetiracetam administration compared with the mean drinks per day consumed during placebo administration.
2. Obtain blood that will be banked for future genetic analysis of polymorphisms in genes that may predict the level of response to alcohol or effects of levetiracetam on alcohol consumption.
3. Test whether the AccuswayTM platform can detect changes in body sway in light to moderate or heavy social drinkers and in subjects taking levetiracetam versus placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults who are social drinkers 21 and 50 years of age.
2. Moderate to heavy social drinkers (women=7-21 drinks/week, men=7-25 drinks/week).
3. Body Mass Index (BMI)>18 and <30.
4. If female, must be non-lactating, not pregnant, and using a reliable contraception method (i.e. abstinence, intrauterine device [IUD], hormonal birth control, or double barrier method [male condom, female condom, or diaphragm plus a spermicidal agent such as contraceptive foam, jelly or cream]).
5. Able and willing to provide written informed consent.
6. Able to understand and follow the instructions of the investigator, and understand all rating scales.
7. Have a negative urine drug screen at all visits, with the exception of cannabinoids.

Exclusion Criteria:

1. Positive urine drug screen, except cannabinoids. Occasional cannabinoid use is allowed, however daily use, dependence, or if considered more than a casual user by study physician, subject will be excluded.
2. Use of cocaine, amphetamines or other stimulants, hallucinogens, ecstasy or other psychoactive drugs, greater than 10 times in the last 24 months or at anytime in the past 60 days.
3. Lifetime use of PCP or ketamine greater than 10 times, or at any time in the last 24 months.
4. History of abusing inhalants (such as glue, toluene or other volatile substances).
5. Current or past dependence on, or addiction to any psychoactive drug (except nicotine or caffeine) including alcohol, as determined by the study physician's assessment.
6. Current or prior enrollment in an alcohol or other drug treatment program, or current legal problems relating to alcohol or other drug use, including awaiting trial or supervision by a parole or probation officer.
7. Binge drinking more than three times per week (binge defined as >5 standard drinks in one session).
8. Alcohol consumption >21 drinks/week for women and >25 drinks/week for men.
9. Currently trying to quit alcohol and/or recreational drug use.
10. Positive for lifetime abnormal opioid use or prescription drug abuse.
11. Clinically significant medical or psychiatric illness (including anxiety or panic disorders) as determined by screening blood tests, medical history, and physical exam performed or reviewed by the study physician.
12. Bilirubin more than 2 times the normal upper limit.
13. AST (SGOT), ALT (SGPT), or alkaline phosphatase more than 2 times the normal upper limit.
14. Body Mass Index >30 or <18
15. Pregnancy or a woman of child bearing potential not currently using an adequate means of contraception.
16. Currently taking any medication other than over-the-counter nonsteroidal anti-inflammatories, acetaminophen, inhaled asthma therapy, contraceptives, nicotine patches, and over-the-counter non-sedating antihistamines.NSAIDs, acetaminophen, or any other OTC (including herbal) medication (unless cleared by study physician).
17. BAC level greater than 0.02% at the beginning of visits 1, 7, or 8 (within margin of error for detection).
18. Estimated creatinine clearance < 50 ml/min.
19. Chronic pain condition requiring regular physician visits and treatment under a physician's supervision.
20. Neurological dysfunction or psychiatric disorder severe enough to interfere with assessment of outcome measures as defined above.
21. Allergy to levetiracetam.
22. Significant cardiac pathology or abnormal initial EKG with QT/QTc interval prolongation > 480 m secs at baseline.
23. Has received an investigational drug within 30 days prior to Study Visit 2 (after screening visit).
24. Subjects who are unable to read or speak English.
25. Those, in the opinion of the investigator, who are considered unable to adhere to scheduled appointments, unlikely to comply with the study protocol, or who are unsuitable for any other reason.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert O. Messing, M.D., Principal Investigator — UCSF; Department of Neurology; Ernest Gallo Clinic and Research Center; Jennifer M. Mitchell, Ph.D., Principal Investigator — UCSF; Department of Neurology; Ernest Gallo Clinic and Research Center
Locations (1):
- Children's Hospital Oakland Research Institute- CRC, Berkeley, California, United States

REFERENCES:
- [Background] Angehagen M, Margineanu DG, Ben-Menachem E, Ronnback L, Hansson E, Klitgaard H. Levetiracetam reduces caffeine-induced Ca2+ transients and epileptiform potentials in hippocampal neurons. Neuroreport. 2003 Mar 3;14(3):471-5. doi: 10.1097/00001756-200303030-00035. PMID 12634506
- [Background] Ardid D, Lamberty Y, Alloui A, Coudore-Civiale MA, Klitgaard H, Eschalier A. Antihyperalgesic effect of levetiracetam in neuropathic pain models in rats. Eur J Pharmacol. 2003 Jul 18;473(1):27-33. doi: 10.1016/s0014-2999(03)01933-2. PMID 12877934
- [Background] Brockmoller J, Thomsen T, Wittstock M, Coupez R, Lochs H, Roots I. Pharmacokinetics of levetiracetam in patients with moderate to severe liver cirrhosis (Child-Pugh classes A, B, and C): characterization by dynamic liver function tests. Clin Pharmacol Ther. 2005 Jun;77(6):529-41. doi: 10.1016/j.clpt.2005.02.003. PMID 15961984
- [Background] Cataldi M, Lariccia V, Secondo A, di Renzo G, Annunziato L. The antiepileptic drug levetiracetam decreases the inositol 1,4,5-trisphosphate-dependent [Ca2+]I increase induced by ATP and bradykinin in PC12 cells. J Pharmacol Exp Ther. 2005 May;313(2):720-30. doi: 10.1124/jpet.104.079327. Epub 2005 Jan 11. PMID 15644427
- [Background] Dong M, Yeh F, Tepp WH, Dean C, Johnson EA, Janz R, Chapman ER. SV2 is the protein receptor for botulinum neurotoxin A. Science. 2006 Apr 28;312(5773):592-6. doi: 10.1126/science.1123654. Epub 2006 Mar 16. PMID 16543415
- [Background] Grunewald R. Levetiracetam in the treatment of idiopathic generalized epilepsies. Epilepsia. 2005;46 Suppl 9:154-60. doi: 10.1111/j.1528-1167.2005.00329.x. PMID 16302890
- [Background] Kim C, Jun K, Lee T, Kim SS, McEnery MW, Chin H, Kim HL, Park JM, Kim DK, Jung SJ, Kim J, Shin HS. Altered nociceptive response in mice deficient in the alpha(1B) subunit of the voltage-dependent calcium channel. Mol Cell Neurosci. 2001 Aug;18(2):235-45. doi: 10.1006/mcne.2001.1013. PMID 11520183
- [Background] Krebs M, Leopold K, Richter C, Kienast T, Hinzpeter A, Heinz A, Schaefer M. Levetiracetam for the treatment of alcohol withdrawal syndrome: an open-label pilot trial. J Clin Psychopharmacol. 2006 Jun;26(3):347-9. doi: 10.1097/01.jcp.0000219926.49799.89. No abstract available. PMID 16702910
- [Background] LaMotte RH, Lundberg LE, Torebjork HE. Pain, hyperalgesia and activity in nociceptive C units in humans after intradermal injection of capsaicin. J Physiol. 1992 Mar;448:749-64. doi: 10.1113/jphysiol.1992.sp019068. PMID 1593488
- [Background] Lipscomb TR, Carpenter JA, Nathan PE. Static ataxia: a predictor of alcoholism? Br J Addict Alcohol Other Drugs. 1979 Sep;74(3):289-94. doi: 10.1111/j.1360-0443.1979.tb01350.x. No abstract available. PMID 290377
- [Background] Lipscomb TR, Nathan PE. Blood alcohol level discrimination. The effects of family history of alcoholism, drinking pattern, and tolerance. Arch Gen Psychiatry. 1980 May;37(5):571-6. doi: 10.1001/archpsyc.1980.01780180085010. PMID 7377914
- [Background] Lukyanetz EA, Shkryl VM, Kostyuk PG. Selective blockade of N-type calcium channels by levetiracetam. Epilepsia. 2002 Jan;43(1):9-18. doi: 10.1046/j.1528-1157.2002.24501.x. PMID 11879381
- [Background] Lynch BA, Lambeng N, Nocka K, Kensel-Hammes P, Bajjalieh SM, Matagne A, Fuks B. The synaptic vesicle protein SV2A is the binding site for the antiepileptic drug levetiracetam. Proc Natl Acad Sci U S A. 2004 Jun 29;101(26):9861-6. doi: 10.1073/pnas.0308208101. Epub 2004 Jun 21. PMID 15210974
- [Background] Madeja M, Margineanu DG, Gorji A, Siep E, Boerrigter P, Klitgaard H, Speckmann EJ. Reduction of voltage-operated potassium currents by levetiracetam: a novel antiepileptic mechanism of action? Neuropharmacology. 2003 Oct;45(5):661-71. doi: 10.1016/s0028-3908(03)00248-x. PMID 12941379
- [Background] Newton PM, Orr CJ, Wallace MJ, Kim C, Shin HS, Messing RO. Deletion of N-type calcium channels alters ethanol reward and reduces ethanol consumption in mice. J Neurosci. 2004 Nov 3;24(44):9862-9. doi: 10.1523/JNEUROSCI.3446-04.2004. PMID 15525770
- [Background] Pisani A, Bonsi P, Martella G, De Persis C, Costa C, Pisani F, Bernardi G, Calabresi P. Intracellular calcium increase in epileptiform activity: modulation by levetiracetam and lamotrigine. Epilepsia. 2004 Jul;45(7):719-28. doi: 10.1111/j.0013-9580.2004.02204.x. PMID 15230693
- [Background] Rigo JM, Hans G, Nguyen L, Rocher V, Belachew S, Malgrange B, Leprince P, Moonen G, Selak I, Matagne A, Klitgaard H. The anti-epileptic drug levetiracetam reverses the inhibition by negative allosteric modulators of neuronal GABA- and glycine-gated currents. Br J Pharmacol. 2002 Jul;136(5):659-72. doi: 10.1038/sj.bjp.0704766. PMID 12086975
- [Background] Rowbotham MC, Manville NS, Ren J. Pilot tolerability and effectiveness study of levetiracetam for postherpetic neuralgia. Neurology. 2003 Sep 23;61(6):866-7. doi: 10.1212/01.wnl.0000079463.16377.07. No abstract available. PMID 14504347
- [Background] Schuckit MA, Smith TL, Kalmijn J. Findings across subgroups regarding the level of response to alcohol as a risk factor for alcohol use disorders: a college population of women and Latinos. Alcohol Clin Exp Res. 2004 Oct;28(10):1499-508. doi: 10.1097/01.alc.0000141814.80716.32. PMID 15597082
- [Background] Saegusa H, Kurihara T, Zong S, Kazuno A, Matsuda Y, Nonaka T, Han W, Toriyama H, Tanabe T. Suppression of inflammatory and neuropathic pain symptoms in mice lacking the N-type Ca2+ channel. EMBO J. 2001 May 15;20(10):2349-56. doi: 10.1093/emboj/20.10.2349. PMID 11350923
- [Result] Hatakeyama S, Wakamori M, Ino M, Miyamoto N, Takahashi E, Yoshinaga T, Sawada K, Imoto K, Tanaka I, Yoshizawa T, Nishizawa Y, Mori Y, Niidome T, Shoji S. Differential nociceptive responses in mice lacking the alpha(1B) subunit of N-type Ca(2+) channels. Neuroreport. 2001 Aug 8;12(11):2423-7. doi: 10.1097/00001756-200108080-00027. PMID 11496122
- [Derived] Mitchell JM, Grossman LE, Coker AR, Messing RO. The anticonvulsant levetiracetam potentiates alcohol consumption in non-treatment seeking alcohol abusers. J Clin Psychopharmacol. 2012 Apr;32(2):269-72. doi: 10.1097/JCP.0b013e318248ba69. PMID 22367657

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted online (Craigslist) and from publicly posted flyers.
Pre-assignment Details: Enrolled participants were excluded prior to medication dosing if blood testing revealed elevated liver enzymes or if urine testing indicated a pregnancy.
Groups:
- Group A: Crossover Between Low Dose Keppra and Placebo: Group A: Twenty moderate to heavy social alcohol users will receive 250 mg of levetiracetam BID (500 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 500 mg of levetiracetam BID (1,000 mg/day) or will receive a double dose of placebo x 7 days. Participants on active drug for the first 14 days then crossed over to placebo after a 10-14 day washout period. Similarly, participants on placebo for the first 14 days then crossed over to active drug after a 10-14 day washout period.
- Group B: Crossover Between High Dose Keppra and Placebo: Group B: Twenty moderate to heavy social alcohol users will receive 500 mg levetiracetam BID (1000 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 1000 mg levetiracetam BID (2,000 mg per day) x 7 days or will receive a double dose of placebo x 7 days. Participants on active drug for the first 14 days then crossed over to placebo after a 10-14 day washout period. Similarly, participants on placebo for the first 14 days then crossed over to active drug after a 10-14 day washout period.
Period: Overall Study
Arm/Group | Group A: Crossover Between Low Dose Keppra and Placebo | Group B: Crossover Between High Dose Keppra and Placebo
Started | 23 | 23
Completed | 23 | 23
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group A: Crossover Between Low Dose Keppra and Placebo: Group A: Twenty moderate to heavy social alcohol users (women 7-20 drinks/week --moderate 7-14 and heavy 15-20 and men 15-25 drinks/week --moderate 7-14 and heavy 15-25 drinks/week) will receive 250 mg of levetiracetam BID (500 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 500 mg of levetiracetam BID (1,000 mg/day) or will receive a double dose of placebo x 7 days. Participants on active drug for the first 14 days then crossed over to placebo after a 10-14 day washout period. Similarly, participants on placebo for the first 14 days then crossed over to active drug after a 10-14 day washout period.
- Group B: Crossover Between High Dose Keppra and Placebo: Group B: Twenty moderate to heavy social alcohol users (women 7-20 drinks/week --moderate 7-14 and heavy 15-20 and men 15-25 drinks/week --moderate 7-14 and heavy 15-25 drinks/week) will receive 500 mg levetiracetam BID (1000 mg/day) or placebo x 7 days and will be titrated to a maximum dose of 1000 mg levetiracetam BID (2,000 mg per day) x 7 days or will receive a double dose of placebo x 7 days.
  Participants on active drug for the first 14 days then crossed over to placebo after a 10-14 day washout period. Similarly, participants on placebo for the first 14 days then crossed over to active drug after a 10-14 day washout period.
- Total: Total of all reporting groups
Arm/Group | Group A: Crossover Between Low Dose Keppra and Placebo | Group B: Crossover Between High Dose Keppra and Placebo | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 23 | 46
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  United States | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Standard Alcoholic Drinks Per Treatment Period
Description: The primary outcome of this study is to determine the effect of levetiracetam on alcohol consumption as measured by change in # of drinks during each treatment period.
Time Frame: During each 14 day treatment period
Population: All study participants were used for data analysis. If there were no significant differences between the two doses of levetiracetam, data would be collapsed for analysis.
Measure: Mean (Standard Error); unit: number of drinks per treatment period
Groups:
- All Subjects (n = 46) Placebo; All Subjects (n = 46) Levetiracetam: 23 moderate social drinkers. 23 heavy social drinkers.
Arm/Group | All Subjects (n = 46) Placebo | All Subjects (n = 46) Levetiracetam
Number analyzed (Participants) | 46 | 46
number of drinks per treatment period | 41.2 (2.8) | 45.4 (3.6)

ADVERSE EVENTS:
Arm/Group | All Subjects (n = 46) Placebo | All Subjects (n = 46) Levetiracetam
Serious Adverse Events (participants affected / at risk) | 0/46 | 0/46
Other Adverse Events (participants affected / at risk) | 0/46 | 0/46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes